CLINICAL TRIAL: NCT05298748
Title: Womb Recordings and Respiratory Control Maturation in Neonates
Brief Title: The Effect of Womb Recordings on Maturation of Respiratory Control in Preterm Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY20211638
Record Dates: First submitted 2022-03-08; First posted 2022-03-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Apnea of Prematurity; Intermittent Hypoxemia; Bradycardia
Keywords: apnea, intermittent hypoxemia, bradycardia, audio recording
MeSH Terms: conditions — Apnea; Bradycardia

STUDY DESIGN:
Intervention Model Description: This is a single site, single visit study. The order of exposure, two 6 hour periods of ambient noise and two 6 hour periods of sound, will be randomized within each subject for a total of 24hrs of sound exposure.
Who Masked: Outcomes Assessor
Masking Description: The order of the sound exposure will be randomized within each subject. The outcomes assessor (quantifying cardiorespiratory events) will be blinded as to the order of the 6 hour randomization blocks within the 24 hour study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambient noise followed by Womb sound (Other): At 34 weeks corrected age, preterm infants (29-33 weeks gestational age at birth), who are off respiratory support >1.5 lpm, will be exposed to alternating 6-hour periods of a recording of ambient noise followed by commercially available womb sounds over a 24-hour period for a combined total of 12 hours of womb sounds and 12 hours of ambient noise.
  Interventions: Other: Womb sound recordings
- Womb sound recordings followed by ambient noise (Other): At 34 weeks corrected age, preterm infants (29-33 weeks gestational age at birth), who are off respiratory support >1.5 lpm, will be exposed to alternating 6-hour periods of a recording of commercially available womb sounds followed by ambient noise over a 24-hour period for a combined total of 12 hours of womb sounds and 12 hours of ambient noise.
  Interventions: Other: Womb sound recordings

INTERVENTIONS:
Other: Womb sound recordings — Womb sounds will be chosen from commercially available (Amazon) womb recordings using a recording that most closely resembles the womb including maternal heart rate, fetal heartbeat, respiratory sounds, bowel "popping" sounds and frequency spectra as described by Parga, Daland 2018 et al.

SUMMARY:
The aim of this proposal is to characterize the acute effect of early postnatal sound exposure on neuronal maturation of the respiratory control regions of the brain in preterm infants.

DETAILED DESCRIPTION:
The aim of this proposal is to characterize the acute effect of early postnatal sound exposure on neuronal maturation of the respiratory control regions of the brain in preterm infants. We hypothesize that exposure to appropriately designed womb-like sounds in the Neonatal Intensive Care Unit (NICU) will induce a more mature and stabilized cardiorespiratory pattern manifesting as a decrease in apnea, bradycardia, intermittent hypoxemia and mean heart rate.

This proposal lays the foundation for further development of actual womb and maternal voice recordings containing components that closely mimic the womb environment during 33-34 weeks of gestation, a proposed therapeutic window of brain development. These sound recordings will provide low risk interventions sorely needed to stabilize respiration, reduce intermittent hypoxemia and induce maturation of neuronal respiratory networks during this critical stage of development.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants 29-33 weeks gestational age at birth
* 34 weeks corrected age
* off respiratory support >1.5 lpm

Exclusion Criteria:

* on respiratory support >1.5 lpm
* congenital anomalies

Ages: 1 Week to 5 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
cardiorespiratory events | During the 24 hour period of randomized blocks of womb sound recordings and ambient noise
  Apnea (>20 seconds or shorter with intermittent hypoxemia <85% or bradycardia <80bpm)
intermittent hypoxemia | During the 24 hour period of randomized blocks of womb sound recordings and ambient noise
  falls in oxygen saturation <85%
mean heart rate | During the 24 hour period of randomized blocks of womb sound recordings and ambient noise
  mean heart rate
bradycardia | During the 24 hour period of randomized blocks of womb sound recordings and ambient noise
  heart rate <80bpm
body motion | During the 24 hour period of randomized blocks of womb sound recordings and ambient noise
  non-cardiac alterations in the oximeter plethysmograph waveform
respiratory pauses | During the 24 hour period of randomized blocks of womb sound recordings and ambient noise
  Respiratory pauses of >5sec will be documented to increase the chance of capturing small alterations in respiratory stability.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Bearer, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noise: a hazard for the fetus and newborn. American Academy of Pediatrics. Committee on Environmental Health. Pediatrics. 1997 Oct;100(4):724-7. No abstract available. PMID 9836852
- [Background] Jobe AH, Bancalari E. An All-Inclusive Perspective on Bronchopulmonary Dysplasia. J Pediatr. 2021 Jul;234:257-259. doi: 10.1016/j.jpeds.2021.03.063. Epub 2021 Apr 1. No abstract available. PMID 33811871
- [Background] White RD, Smith JA, Shepley MM; Committee to Establish Recommended Standards for Newborn ICU Design. Recommended standards for newborn ICU design, eighth edition. J Perinatol. 2013 Apr;33 Suppl 1:S2-16. doi: 10.1038/jp.2013.10. PMID 23536026
- [Result] Almadhoob A, Ohlsson A. Sound reduction management in the neonatal intensive care unit for preterm or very low birth weight infants. Cochrane Database Syst Rev. 2015 Jan 30;1:CD010333. doi: 10.1002/14651858.CD010333.pub2. PMID 25633155
- [Result] Barateiro A, Brites D, Fernandes A. Oligodendrocyte Development and Myelination in Neurodevelopment: Molecular Mechanisms in Health and Disease. Curr Pharm Des. 2016;22(6):656-79. doi: 10.2174/1381612822666151204000636. PMID 26635271
- [Result] Benzaquen S, Gagnon R, Hunse C, Foreman J. The intrauterine sound environment of the human fetus during labor. Am J Obstet Gynecol. 1990 Aug;163(2):484-90. doi: 10.1016/0002-9378(90)91180-k. PMID 2386134
- [Result] Brockmann PE, Wiechers C, Pantalitschka T, Diebold J, Vagedes J, Poets CF. Under-recognition of alarms in a neonatal intensive care unit. Arch Dis Child Fetal Neonatal Ed. 2013 Nov;98(6):F524-7. doi: 10.1136/archdischild-2012-303369. Epub 2013 May 28. PMID 23716498
- [Result] Coleman RJ, Beharry KD, Brock RS, Abad-Santos P, Abad-Santos M, Modanlou HD. Effects of brief, clustered versus dispersed hypoxic episodes on systemic and ocular growth factors in a rat model of oxygen-induced retinopathy. Pediatr Res. 2008 Jul;64(1):50-5. doi: 10.1203/PDR.0b013e31817307ac. PMID 18344903
- [Result] Corrigan MJ, Keeler JR, Miller HD, Ben Khallouq BA, Fowler SB. Music therapy and retinopathy of prematurity screening: using recorded maternal singing and heartbeat for post exam recovery. J Perinatol. 2020 Dec;40(12):1780-1788. doi: 10.1038/s41372-020-0719-9. Epub 2020 Jul 17. PMID 32681063
- [Result] Decker MJ, Rye DB. Neonatal intermittent hypoxia impairs dopamine signaling and executive functioning. Sleep Breath. 2002 Dec;6(4):205-10. doi: 10.1007/s11325-002-0205-y. PMID 12524574
- [Result] Di Fiore JM, Bloom JN, Orge F, Schutt A, Schluchter M, Cheruvu VK, Walsh M, Finer N, Martin RJ. A higher incidence of intermittent hypoxemic episodes is associated with severe retinopathy of prematurity. J Pediatr. 2010 Jul;157(1):69-73. doi: 10.1016/j.jpeds.2010.01.046. Epub 2010 Mar 20. PMID 20304417
- [Result] Di Fiore JM, Kaffashi F, Loparo K, Sattar A, Schluchter M, Foglyano R, Martin RJ, Wilson CG. The relationship between patterns of intermittent hypoxia and retinopathy of prematurity in preterm infants. Pediatr Res. 2012 Dec;72(6):606-12. doi: 10.1038/pr.2012.132. Epub 2012 Oct 4. PMID 23037873
- [Result] Doheny L, Hurwitz S, Insoft R, Ringer S, Lahav A. Exposure to biological maternal sounds improves cardiorespiratory regulation in extremely preterm infants. J Matern Fetal Neonatal Med. 2012 Sep;25(9):1591-4. doi: 10.3109/14767058.2011.648237. Epub 2012 Feb 2. PMID 22185623
- [Result] Emery L, Hamm EL, Hague K, Chorna OD, Moore-Clingenpeel M, Maitre NL. A randomised controlled trial of protocolised music therapy demonstrates developmental milestone acquisition in hospitalised infants. Acta Paediatr. 2019 May;108(5):828-834. doi: 10.1111/apa.14628. Epub 2018 Dec 7. PMID 30375661
- [Result] Jiang NM, Cowan M, Moonah SN, Petri WA Jr. The Impact of Systemic Inflammation on Neurodevelopment. Trends Mol Med. 2018 Sep;24(9):794-804. doi: 10.1016/j.molmed.2018.06.008. Epub 2018 Jul 11. PMID 30006148
- [Result] Jobe AH, Kallapur SG. Long term consequences of oxygen therapy in the neonatal period. Semin Fetal Neonatal Med. 2010 Aug;15(4):230-5. doi: 10.1016/j.siny.2010.03.007. Epub 2010 May 10. PMID 20452844
- [Result] Lahav A, Skoe E. An acoustic gap between the NICU and womb: a potential risk for compromised neuroplasticity of the auditory system in preterm infants. Front Neurosci. 2014 Dec 5;8:381. doi: 10.3389/fnins.2014.00381. eCollection 2014. PMID 25538543
- [Result] Loewy J, Stewart K, Dassler AM, Telsey A, Homel P. The effects of music therapy on vital signs, feeding, and sleep in premature infants. Pediatrics. 2013 May;131(5):902-18. doi: 10.1542/peds.2012-1367. Epub 2013 Apr 15. PMID 23589814
- [Result] Parga JJ, Bhatt RR, Kesavan K, Sim MS, Karp HN, Harper RM, Zeltzer L. A prospective observational cohort study of exposure to womb-like sounds to stabilize breathing and cardiovascular patterns in preterm neonates. J Matern Fetal Neonatal Med. 2018 Sep;31(17):2245-2251. doi: 10.1080/14767058.2017.1339269. Epub 2017 Jun 22. PMID 28587528
- [Result] Parga JJ, Daland R, Kesavan K, Macey PM, Zeltzer L, Harper RM. A description of externally recorded womb sounds in human subjects during gestation. PLoS One. 2018 May 10;13(5):e0197045. doi: 10.1371/journal.pone.0197045. eCollection 2018. PMID 29746604
- [Result] Peng YJ, Prabhakar NR. Effect of two paradigms of chronic intermittent hypoxia on carotid body sensory activity. J Appl Physiol (1985). 2004 Mar;96(3):1236-42; discussion 1196. doi: 10.1152/japplphysiol.00820.2003. Epub 2003 Dec 5. PMID 14660510
- [Result] Poets CF, Roberts RS, Schmidt B, Whyte RK, Asztalos EV, Bader D, Bairam A, Moddemann D, Peliowski A, Rabi Y, Solimano A, Nelson H; Canadian Oxygen Trial Investigators. Association Between Intermittent Hypoxemia or Bradycardia and Late Death or Disability in Extremely Preterm Infants. JAMA. 2015 Aug 11;314(6):595-603. doi: 10.1001/jama.2015.8841. PMID 26262797
- [Result] Raffaeli G, Manzoni F, Cortesi V, Cavallaro G, Mosca F, Ghirardello S. Iron Homeostasis Disruption and Oxidative Stress in Preterm Newborns. Nutrients. 2020 May 27;12(6):1554. doi: 10.3390/nu12061554. PMID 32471148
- [Result] Raffay TM, Dylag AM, Sattar A, Abu Jawdeh EG, Cao S, Pax BM, Loparo KA, Martin RJ, Di Fiore JM. Neonatal intermittent hypoxemia events are associated with diagnosis of bronchopulmonary dysplasia at 36 weeks postmenstrual age. Pediatr Res. 2019 Feb;85(3):318-323. doi: 10.1038/s41390-018-0253-z. Epub 2018 Dec 12. PMID 30538265
- [Result] Rains ME, Muncie CB, Pang Y, Fan LW, Tien LT, Ojeda NB. Oxidative Stress and Neurodevelopmental Outcomes in Rat Offspring with Intrauterine Growth Restriction Induced by Reduced Uterine Perfusion. Brain Sci. 2021 Jan 8;11(1):78. doi: 10.3390/brainsci11010078. PMID 33435577
- [Result] Reeves SR, Gozal D. Developmental plasticity of respiratory control following intermittent hypoxia. Respir Physiol Neurobiol. 2005 Nov 15;149(1-3):301-11. doi: 10.1016/j.resp.2005.01.014. PMID 16203218
- [Result] Reeves SR, Mitchell GS, Gozal D. Early postnatal chronic intermittent hypoxia modifies hypoxic respiratory responses and long-term phrenic facilitation in adult rats. Am J Physiol Regul Integr Comp Physiol. 2006 Jun;290(6):R1664-71. doi: 10.1152/ajpregu.00851.2005. Epub 2006 Feb 2. PMID 16455761
- [Result] Smith CV, Satt B, Phelan JP, Paul RH. Intrauterine sound levels: intrapartum assessment with an intrauterine microphone. Am J Perinatol. 1990 Oct;7(4):312-5. doi: 10.1055/s-2007-999511. PMID 2222618
- [Result] Smith SW, Ortmann AJ, Clark WW. Noise in the neonatal intensive care unit: a new approach to examining acoustic events. Noise Health. 2018 Jul-Aug;20(95):121-130. doi: 10.4103/nah.NAH_53_17. PMID 30136672
- [Result] Standley J. Music therapy research in the NICU: an updated meta-analysis. Neonatal Netw. 2012 Sep-Oct;31(5):311-6. doi: 10.1891/0730-0832.31.5.311. PMID 22908052
- [Result] Stokes A, Agthe AG, El Metwally D. Music exposure and maturation of late preterm sleep-wake cycles: a randomised crossover trial. Acta Paediatr. 2018 Apr;107(4):582-586. doi: 10.1111/apa.14079. Epub 2017 Oct 11. PMID 28929527
- [Result] Volpe JJ. Brain injury in premature infants: a complex amalgam of destructive and developmental disturbances. Lancet Neurol. 2009 Jan;8(1):110-24. doi: 10.1016/S1474-4422(08)70294-1. PMID 19081519